CLINICAL TRIAL: NCT04891276
Title: Impact of COVID-19 Infection and Confinement on Diabetic Ulcer Management and Amputation Risk
Acronym: COROPIEDIAB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: PETIT SERI 2020
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Subjects With Hospital Stays
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data collection on the national PMSI database

SUMMARY:
In the context of the COVID-19 pandemic, a number of factors, including the lockdown that was imposed to limit the spread of infection, the fear of being contaminated during hospital consultations and the difficulty in accessing general practitioners may have led to delays in the referral of patients to facilities specialized in the management of diabetic ulcers. Since the beginning of the coronavirus pandemic and during the first lockdown, we observed a clear decrease in hospitalizations and consultations for diabetic ulcers. Patients who had regular follow-up for the management of their diabetic ulcers cancelled their scheduled appointments for fear of being contaminated in the hospital. It is feared that the current epidemic context has favored the delay of referral of patients with diabetic ulcers to specialized facilities, with consequences on the prognosis of these patients and the risk of lower limb amputation.

In this context, this project aims to evaluate the impact of confinement on emergency hospitalizations for foot wounds and the effects on the risk of amputation during the lockdown and the three months following the end of the lockdown.

Our hypothesis is that the lockdown led to a decrease in hospitalizations for foot wounds, resulting in a delay in the management of these patients, and potentially leading to an increase in the number of amputations in the three months following the end of the lockdown.

In parallel, we will also study the impact of confinement on deferrable hospitalizations (glycemic imbalance, assessment of diabetic complications...) or theoretically non-deferrable (diabetic comas, ketoacidosis, diagnosis of type 1 diabetes, acute coronary syndrome, stroke...) of diabetes mellitus. This will allow us to evaluate whether our findings relative to diabetic ulcers could be extended to other complications of diabetes.

ELIGIBILITY:
Inclusion Criteria:

Diabetic subjects with hospital stays in France, 2017 to 2020.

Exclusion Criteria:

Absence of diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetic subjects with hospital stays in France, 2017 to 2020.
Sampling Method: Non-Probability Sample
Enrollment: 3300000 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Frequency of lower limb amputations | 3 months after the end of the spring 2020 lockdown

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Mariet AS, Benzenine E, Bouillet B, Verges B, Quantin C, Petit JM. Impact of the COVID-19 Epidemic on hospitalization for diabetic foot ulcers during lockdown: A French nationwide population-based study. Diabet Med. 2021 Jul;38(7):e14577. doi: 10.1111/dme.14577. Epub 2021 Apr 13. PMID 33797791